CLINICAL TRIAL: NCT03543345
Title: The Changes in The Right Ventricular Function After Elective Percutaneous Coronary Intervention in Patients With Right Coronary Artery Occlusion
Brief Title: Right Ventricular Function Change After PCI to Right Coronary Artery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hazim Alaa, Principal investigator, Assiut University
Other Study IDs: HAZ190
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Right Coronary Artery Occlusion
Keywords: RCA; PCI; right ventricular function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: echocardiography study — Patients with right coronary artery occlusion lesion will be subjected to:
  * Written consent.
  * Complete history.
  * Complete physical examination.
  * Trans-thoracic echocardiography assessment of the right ventricular function before PCI to the RCA
  * Follow up Trans-thoracic echocardiography assessment of the right ventricular function four weeks after the PCI.

SUMMARY:
Proximal RCA occlusions were very often found among men with fatal pre-hospital MI; whereas left-sided coronary occlusions were significantly more frequent in hospital-admitted survivors of MI. Left-sided coronary occlusions may be associated with a more favorable pre-hospital phase of acute MI compared to proximal RCA occlusions. Proximal RCA occlusion increases the risk of arrhythmia and shock leading to increase the mortality. Sinus bradycardia and cardiogenic shock accounts for the majorities of the mortalities of RCA occlusion

DETAILED DESCRIPTION:
Myocardial infarction is a common presentation of coronary artery disease. The World Health Organization estimated in 2004, that 12.2% of worldwide deaths were from ischemic heart disease; with it being the leading cause of death in high- or middle-income countries and second only to lower respiratory infections in lower-income countries. Worldwide, more than 3 million people have STEMIs and 4 million have NSTEMIs a year . STEMIs occur about twice as often in men as women .

Myocardial infarction means that the tissue ischemia caused tissue death, as a result of diminished blood supply to a part of the heart muscles. The blood supply of the heart is coronary arteries (right and left). Proximal RCA occlusions were very often found among men with fatal pre-hospital MI; whereas left-sided coronary occlusions were significantly more frequent in hospital-admitted survivors of MI. Left-sided coronary occlusions may be associated with a more favorable pre-hospital phase of acute MI compared to proximal RCA occlusions .

The right coronary artery (RCA) supplies the right ventricle, 25% to 35% of the left ventricle and SA node in 60% of people. Proximal RCA occlusion increases the risk of arrhythmia and shock leading to increase the mortality. Sinus bradycardia and cardiogenic shock accounts for the majorities of the mortalities of RCA occlusion.

Sinus bradycardia is more frequent when the infarct-related artery is the RCA than other arteries involvement. Proximal occlusions of the RCA presented sinus bradycardia more than medial and distal occlusions.

Mortality of cardiogenic shock due to right ventricular infarction (55%) was comparable to that due to left ventricular infarction (59%) in spite of patients being younger and a greater incidence of single vessel disease. The worse prognosis in patients with RV myocardial involvement may be related to the increased risk of life-threatening ventricular arrhythmias in these patients.

Approximately one half of patients who present with signs and symptoms of acute inferior myocardial infarction have proximal occlusion of the dominant right coronary artery (RCA) and also show ECG signs of RV wall ischemia or infarction. Occlusion sufficiently proximal to cause RV free wall injury also frequently compromises the blood supply to the sinoatrial node, atrium and atrioventricular (AV) node, producing such effects as sinus bradycardia, atrial infarction, atrial fibrillation and AV block.

The transthoracic echocardiography is the most common method to assess the function of the right ventricular function as it non-invasive, inexpensive and available in most of the hospitals. The presence of RV dysfunction on early echocardiography is an important predictor of an adverse prognosis, both short-and long-term, in STEMI patients.

The Tissue Doppler Imaging method depicts myocardial motion (measured as tissue velocity) at specific locations in the heart. Tissue velocity indicates the rate at which a particular point in the myocardium moves toward or away from the transducer. Integration of velocity over time yields displacement or the absolute distance moved by that point.

Evaluation of right ventricular function by echocardiography is challenging and often ignored in clinical practice. Tricuspid annular velocity correlates with right ventricular ejection fraction . Tricuspid annular excursion (tricuspid displacement) predicted 2-year survival in patients with pulmonary hypertension . Isovolumic acceleration, derived from tissue velocity, is a load-independent measure of contractility and correlates with right ventricular end-systolic elastance. This correlation is less pronounced in clinical studies . More recent experimental data suggest a weak relationship between isovolumic acceleration and regional contractility. Systolic velocity and strain best correlated with invasively determined right ventricular stroke volume and dynamically tracked changes in right ventricular function during vasodilator infusion. Strain rates and strain quantitate regional right ventricular systolic function in various pathologies

ELIGIBILITY:
Inclusion Criteria:

* Patients subjected to elective PCI due to right coronary artery occlusion. Patients between 40 and 75 years old from the both genders

Exclusion Criteria:

1. History of chronic respiratory condition and PHTN
2. Patients with previous percutaneous coronary intervention (PCI) or coronary artery bypass graft surgery (CABG).
3. History of valvular surgery.
4. Patients with significant rheumatic vavular heart disease.
5. Presence of persistant arrythemia
6. Patients with End stage renal disease.
7. Patients with End stage liver disease.
8. Haemodynamically unstable patients.
9. Patients with previous Myocardial infarction.
10. Patients with Ischemic Dilated Cardiomyopathy.
11. Patients with pericardial disease.
12. Patients with congenital intra-cardiac shunt.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients subjected to elective PCI due to right coronary artery occlusion. Patients between 40 and 75 years old from the both genders
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-08-15 (Estimated); Study Completion 2018-08-28 (Estimated)

PRIMARY OUTCOMES:
Change in RV function PCI to RCA | 3 months
  The aim of the study is to determine the impact of elective PCI of RCA on RV systolic and diastolic functions.

CONTACTS AND LOCATIONS:
Locations (1):
- Al Azhar university, Asyut, Egypt